CLINICAL TRIAL: NCT05898906
Title: Turkish Adaptation, Validity and Reliability Study of Activities Scales for Kids
Brief Title: Turkish Version of the Activity Scales for Kids
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Ozgun Kaya Kara, Assoc. Prof. PhD, Akdeniz University
Other Study IDs: 2022-189
Record Dates: First submitted 2023-06-02; First posted 2023-06-12 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Neurodevelopmental Disorders
Keywords: Activities; Participation; Children
MeSH Terms: conditions — Neurodevelopmental Disorders; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children with special needs Group: Children who have diagnosed neurodevelopment disorders including cerebral palsy, autism spectrum disorder,
- Control Group: Typically developing children

SUMMARY:
Children's participation in age-appropriate activities is critical to their overall well-being. Neurodevelopmental disorders cause motor, cognitive, communication, and behavioural problems. Children have restrictions in their ability to participate and engage in activities because of these problems. Children with neurodevelopmental disorders require more parental care and are less likely to participate in activities at home, school, and in the community than their healthy peers. This highlights the significance of evaluating activity restrictions and participation limitations. Our study aims to demonstrate the reliability and validity of the Turkish version of the Activity Scales for Kids (ASK), which assesses children's participation and activity in their daily lives at home, school, and play, as well as cultural sensitivity.

DETAILED DESCRIPTION:
Participation in activities is an essential component of maintaining health. The International Classification of Functioning- Child and Youth (ICF-CY) framework includes several components that can be used to determine activity and participation. These components are defined by two terms: capacity and performance. Both capacity and performance are basically measures of capability, even if the performance qualifier is intended as a measure of participation. Performance describes what a person does in their current setting. The current environment brings with it a social context. As a result, performance determines how involved an individual is in his or her living environment and life experience. The ability to do a task or action is known as capacity, which denotes the highest functional level that may be achieved at any moment and in every setting. Capacity is measured in a consistent or standard setting. Therefore, it reflects the individually adjusted ability of the individual. The child's physical and social environment has an impact on their capacity. For instance, while the child can stand up on his own in a standardized clinical setting, he might not be able to do the same after falling during physical exercise in a school context or in public.

According to the ICF-CY, disability is not only related to body structure and function but also to activity constraints and participation restrictions in various situations. An objective assessment demonstrates how performance has changed over time and encourages children to enhance their own abilities. These examinations need to meet psychometric standards before being used with children. In addition, the results of research studies provide useful information about the natural developmental steps expected, especially in childhood disability subgroups. There isn't a valid and reliable scale in Turkish literature that assesses children's capacity and performance in activities at home, school, and in play environments. The goals of our research are to demonstrate the reliability and validity of the ASK, a tool that assesses children's participation and activity levels at play, school, and at home. Families and medical professionals will be guided by this scale.

ELIGIBILITY:
Inclusion Criteria:

* Age between 5 years and 15 years;
* Diagnosed with neurodevelopmental disorders.
* To have the cognitive ability to answer questions for assessment.
* Completing the test-retest assessment.
* To be able to read and speak Turkish

Exclusion Criteria:

* Patients with unmanageable psychological disorders (schizophrenia, bipolar disorder, major depressive disorder) would be excluded from the study.

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: children who have diagnosed neurodevelopment disorders
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-07-20 (Estimated); Primary Completion 2023-09-20 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Activities Scales for Kids | Baseline
  The Activities Scales for Kids scale measures pediatric functionality from the perspective of the children. These are ASK-Performance (ASKp) and ASK-Capacity (ASKc). ach version consists of 30 items, including personal care (3 items), dressing (4 items), other skills (4 items), locomotion (7 items), play (2 items), standing (5 items), and transfers (5 items). ASKc evaluates what the child "can do", and ASKp evaluates what the child "usually does". A percentage score (with a range of 0-100) is calculated by dividing this average by 4. On this scale, 100% indicates full physical function.

SECONDARY OUTCOMES:
Participation and Environment- Children and Youth | Baseline
  The participation sections included 10 activities in the home setting, five activities in the school setting, and 10 in the community setting. For each activity, the range of participation is daily to never, with scores between 0 and 8; higher scores indicate greater participation. The range of involvement is from very involved to minimally involved, with scores between 1 and 5; higher scores indicate greater involvement. The range of whether change is desired in the child's participation in this kind of activity is no or yes, with scores between 0 and 1. Environmental features supports and barriers (e.g., do the features of the environment help or make it harder?) for the child to participate in activities at home, school, or in a community setting with scores between 1 and 4; increased scores indicate environmental help.

CONTACTS AND LOCATIONS:
Overall Officials: Ozgun Kaya Kara, Assoc. Prof., Principal Investigator — Akdeniz University
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

REFERENCES:
- [Background] Young NL, Williams JI, Yoshida KK, Wright JG. Measurement properties of the activities scale for kids. J Clin Epidemiol. 2000 Feb;53(2):125-37. doi: 10.1016/s0895-4356(99)00113-4. PMID 10729684
- [Background] Santamaria-Vazquez M, Guijo-Blanco V, Puente-Martinez A, Ubillos-Landa S. Psychometric properties of the Spanish version of the Activities Scale for Kids (ASK): reliability, validity and the Rasch model. BMJ Open. 2023 Apr 27;13(4):e069248. doi: 10.1136/bmjopen-2022-069248. PMID 37105695
- [Background] de Oliveira VGC, Balau LC, Arrebola LS, Young NL, Yi LC. Translation, cross-cultural adaptation, validity and reliability of the Brazilian Portuguese version of Activity Scale for Kids questionnaire. Child Care Health Dev. 2023 Jul;49(4):725-731. doi: 10.1111/cch.13085. Epub 2022 Dec 8. PMID 36444144
- [Background] Shakya R, Suwal R, Adhikari I, Shrestha J, Gyawali S, Shrestha A. Cross cultural adaptation and validation of Nepali Version of Activity Scale for Kids (ASK). J Patient Rep Outcomes. 2022 Jun 16;6(1):68. doi: 10.1186/s41687-022-00479-2. PMID 35708828
- [Background] Fabbri L, Neviani R, Festini F, Costi S. Transcultural validation of Activities Scale for Kids (ASK): translation and pilot test. Acta Biomed. 2016 May 26;87 Suppl 2:70-9. PMID 27240035
- [Background] Paixao D, Cavalheiro LM, Goncalves RS, Ferreira PL. Portuguese cultural adaptation and validation of the Activities Scale for Kids (ASK). J Pediatr (Rio J). 2016 Jul-Aug;92(4):367-73. doi: 10.1016/j.jped.2015.09.010. Epub 2016 May 3. PMID 27151375
- [Background] Costi S, Mecugni D, Beccani L, Alboresi S, Bressi B, Paltrinieri S, Ferrari A, Pelosin E. Construct Validity of the Activities Scale for Kids Performance in Children with Cerebral Palsy: Brief Report. Dev Neurorehabil. 2020 Oct;23(7):474-477. doi: 10.1080/17518423.2020.1764649. Epub 2020 Jun 7. PMID 32508188
- [Background] Kaya Kara O, Turker D, Kara K, Yardimci-Lokmanoglu BN. Psychometric properties of the Turkish version of Participation and Environment Measure for Children and Youth. Child Care Health Dev. 2020 Nov;46(6):711-722. doi: 10.1111/cch.12801. Epub 2020 Aug 19. PMID 32776565
- [Background] Costi S, Filippi MC, Braglia L, Beccani L, Corradi I, Bruzzi E, Signorelli C, Pelosin E. Reliability and construct validity of the Activities Scale for Kids in Italian children with cerebral palsy. Disabil Rehabil. 2022 Oct;44(21):6445-6451. doi: 10.1080/09638288.2021.1966519. Epub 2021 Aug 20. PMID 34415225